CLINICAL TRIAL: NCT00477763
Title: Oasys vs. Extreme H20 Xtra 59
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: Thomas Kislan, OD, Hazleton Eye Specialists
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 5300
Record Dates: First submitted 2007-05-21; First posted 2007-05-24 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Restasis, Refresh Endura
- 2 (Placebo Comparator)
  Interventions: Drug: Restasis, Refresh Endura

INTERVENTIONS:
Drug: Restasis, Refresh Endura — 1. Restasis 0.4ml- (in the eye) instill twice daily in the randomized eye morning and evening
  2. Refresh Endura 0.4ml- (in the eye) instill twice daily in the randomized eye morning and evening

SUMMARY:
To compare the performance of Oasys to Extreme H20 xtra 59 in dry eye contact lens pts who receive Restasis in 1 eye and vehicle (Endura) in the other eye.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 19 years of age
* Contact Lens Wearers
* Patients with mild to moderate symptoms of dry eye

Exclusion Criteria:

* male or female younger than 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
comparing performance of contact lens | 10 months

SECONDARY OUTCOMES:
Dry eye | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kislan, OD, Principal Investigator — Hazleton Eye Specialists
Locations (1):
- Hazleton Eye Specialists, Hazleton, Pennsylvania, United States